CLINICAL TRIAL: NCT02368782
Title: Effects of Ketamine and Propofol in Otoacoustic Emissions (OAE) in Children With Normal Hearing Tests Undergoing Adenoidectomy and Tonsillectomy
Brief Title: Effects of Ketamine and Propofol in Otoacoustic Emissions (OAE) in Children
Acronym: OAE
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Prof. Dr. A. Pervin SUTAS BOZKURT, Prof. Dr., Istanbul University
Other Study IDs: 30112011; 36171 (Other Grant/Funding Number: ıstanbul University Scientific Research Department)
Record Dates: First submitted 2014-08-27; First posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Normal Healthy Ears; Ketamine and Propofol Effects on Hemodynamics; Ketamine and Propofol Effects on TEOAE and DPOAE
Keywords: transient evoked otoacoustic emissions; distortion product otoacoustic emissions; ketamine; propofol; child

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ketamine group: ketamine 2mg/kg bolus IV once
- propofol group: propofol 2mg/kg ıv bolus once

SUMMARY:
Otoacoustic emissions (OAEs) are non-invasive, easy to apply and objective test methods which are widely used to determine the presence of hearing in audiology clinics. Under some circumstances and children, the study should be applied under general anaesthesia. The aim of this study was to find out the influence of propofol (P) and ketamine (K) on OAE measurements. .

Methods: Thirty- healthy children who will underwent adenoidectomy and tonsillectomy will be included in this study after Institutional ethics committee approval and informed consent of parents. Children will be evaluated one day before surgery by tympanometry. Psychologically prepared children will be admitted to the operating room. Following EMLA (Eutectic Mixture of Local Anesthetics ) cream application IV line will be inserted. ECG and non-invasive blood pressure will be monitored. Transient evoked otoacoustic emissions (TEOAEs) and distortion product otoacoustic emissions (DPOAEs) will measured in both ears of each patient (n=20 ears) prior to P or K administration( Pre-P and Pre-K). Propofol will be given 2mg/kg or ketamine 2mg/kg intravenously and 40% O2 in air will be given by mask ventilation. Five minutes later TEOAE and DPOAE measurements will be repeated (Post-P and Post-K). After this measurement the routine general anaesthesia and surgical protocol will be commenced. Heart rate, blood pressures TEOAE and DPOAE measurements will be compared at pre and post stages by paired Student's t- test.

ELIGIBILITY:
Inclusion Criteria:

children ages 4-15 years ASA ( American Society of Anesthesiologists) I-II Tonsillectomy and/or adenoidectomy Normal ear hearing tests

Exclusion Criteria:

Abnormal hearing tests Abnormal laboratory (Electrolyte imbalance, anemia, polycythemia, thrombocytopenia, leucopenia , leucocytosis) Congenital abnormalities and previous systemic diseases Hypo or hyperthermia Ear operations Long term fasting, dehydration or over hydration Upper respiratory disease, acute or chronic otitis,

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children ages 4-15 years ASA I-II Tonsillectomy and/or adenoidectomy Normal ear hearing tests
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
DPOAE and TEOAE | Pre and post propofol or ketamine administration
  Before and after the administration of propofol or ketamine measurements of DPOAE and TEOAE will be performed

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Cerrahpasa Medical Faculty, Istanbul, Turkey (Türkiye)